CLINICAL TRIAL: NCT03769545
Title: Mortality Post-TAVI and Correlation With Haemodynamic Parameters.
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Panagiotis Savvoulidis, Clinical Fellow in Interventional Cardiology, Royal Brompton & Harefield NHS Foundation Trust
Other Study IDs: 258843
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Until a few years ago the only interventional option available for severe aortic stenosis was surgical aortic valve replacement. About a decade ago, a novel percutaneous technique was applied for the first time in humans, the transcatheter aortic valve implantation (TAVI). Initially this procedure was reserved for those patients deemed too high risk for surgical intervention. As technology progressed in this domain, the indication for TAVI expanded to a broader population of patient with severe aortic stenosis. To-date there are no long-term data for mortality and this is the central question this study will explore in correlation with haemodynamic parameters. Essentially, this study will explore the effect of TAVI in the long term. All patients that had a TAVI within the RBH&HH NHS Foundation Trust between January 2008 and December 2017 will be included in the study. This is a retrospective study.

DETAILED DESCRIPTION:
Aortic valve stenosis is the most prevalent valvulopathy in the developed world countries. Until a few years ago the only interventional option available for severe aortic stenosis was surgical aortic valve replacement. About a decade ago, a novel percutaneous technique was applied for the first time in humans, the transcatheter aortic valve implantation (TAVI) as a keyhole procedure. Initially this procedure was reserved for those patients deemed too high risk for surgical intervention. As technology progressed in this domain, the indication for TAVI expanded to a broader population of patient with severe aortic stenosis. As the experience broadens there are no long-term data for mortality and this is the central question this study will explore in correlation with haemodynamic parameters. Essentially, this study will explore the effect of TAVI in the long term. All patients that had a TAVI within the RBH&HH NHS Foundation Trust between January 2008 and December 2017 will be included in the study. This is a retrospective study and will not change anything in the patients' standard of care.

ELIGIBILITY:
Inclusion Criteria:

* All patients with TAVI within the Royal Brompton & Harefield NHS Foundation Trust

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with TAVI within the Royal Brompton & Harefield NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Death post-TAVI | Within 3 years from TAVI procedure
  Death during or after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Luescher, Study Director — Director of Research Education and Development, Cardiology (RBH)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Denegri A, Mehran R, Holy E, Taramasso M, Pasotti E, Pedrazzini G, Moccetti T, Maisano F, Nietlispach F, Obeid S. Post procedural risk assessment in patients undergoing trans aortic valve implantation according to the age, creatinine, and ejection fraction-7 score: Advantages of age, creatinine, and ejection fraction-7 in stratification of post-procedural outcome. Catheter Cardiovasc Interv. 2019 Jan 1;93(1):141-148. doi: 10.1002/ccd.27806. Epub 2018 Sep 30. PMID 30269398
- [Background] Cocchieri R, Petzina R, Romano M, Jagielak D, Bonaros N, Aiello M, Lapeze J, Laine M, Chocron S, Muir D, Eichinger W, Thielmann M, Labrousse L, Rein KA, Verhoye JP, Gerosa G, Bapat V, Baumbach H, Sims H, Deutsch C, Bramlage P, Kurucova J, Thoenes M, Frank D. Outcomes after transaortic transcatheter aortic valve implantation: long-term findings from the European ROUTEdagger. Eur J Cardiothorac Surg. 2019 Apr 1;55(4):737-743. doi: 10.1093/ejcts/ezy333. PMID 30346515
- [Background] Adams HSL, Ashokkumar S, Newcomb A, MacIsaac AI, Whitbourn RJ, Palmer S. Contemporary review of severe aortic stenosis. Intern Med J. 2019 Mar;49(3):297-305. doi: 10.1111/imj.14071. PMID 30091235